CLINICAL TRIAL: NCT01847508
Title: A Multicenter Randomized Controlled Trial to Investigate the Treatment Outcome of PHILOS Screw Augmentation Compared to PHILOS Without Augmentation in Older Adult Patients With Proximal Humerus Fractures
Brief Title: PHILOS Augmented - a Multicenter Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHILOS+
Record Dates: First submitted 2013-04-26; First posted 2013-05-07 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Humerus Fractures; Closed Fracture of the Proximal Humerus
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHILOS + (Active Comparator): Proximal Humeral Internal Locking System with screw tip augmentation (PHILOS+) with high viscous polymethylmethacrylate (PMMA) cement (Traumacem V+).
  Interventions: Device: PHILOS+
- PHILOS (Active Comparator): Proximal Humeral Internal Locking System (PHILOS)
  Interventions: Device: PHILOS

INTERVENTIONS:
Device: PHILOS+ — Proximal Humerus Internal Locking System with screw tip augmentation (PHILOS+) with high viscous polymethylmethacrylate (PMMA) cement (Traumacem V+).
  Other Names: PHILOS Length 90 mm with 3 shaft holes; PHILOS Length 114 mm with 5 shaft holes
  Arms: PHILOS +
Device: PHILOS — Proximal Humerus Internal Locking System (PHILOS).
  Other Names: PHILOS Length 90 mm with 3 shaft holes; PHILOS Length 114 mm with 5 shaft holes
  Arms: PHILOS

SUMMARY:
The primary objective is to compare the mechanical failure risks in the first year after treatment.

DETAILED DESCRIPTION:
Biomechanical tests have shown that augmentation of screws or nails with polymethylmethacrylate (PMMA) leads to increased mechanical properties of the bone-implant complex, leading to the assumption that augmentation could reduce mechanical failures in patients. While a few clinical studies have already been performed with augmented trochanteric nails in proximal femur fractures, no clinical studies exist with the use of Proximal Humerus Internal Locking System (PHILOS) and (PMMA) augmentation for the treatment of fractures in the proximal humerus.

In this study a new standardized technique for augmentation of screw tips using high viscous PMMA cement (Traumacem V+) with the PHILOS plate will be applied. Fracture treatment with PHILOS Screw Augmentation will be compared with treatment with PHILOS without augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Low energy trauma (e.g. fall from standing height)
* Radiologically confirmed closed fracture (≤ 10 days) of the proximal humerus
* Any displaced or unstable 3- or 4-part fracture of the proximal humerus (i.e. segment dis-placement > 0.5 cm or angulated > 45°) except isolated displaced fractures of the greater or lesser tuberosity
* Primary fracture treatment with a PHILOS plate
* Ability to understand the content of the patient information / informed consent form
* Willingness and ability to participate in the clinical investigation including imaging and fol-low-up procedures
* Signed informed consent

Preoperative Exclusion Criteria:

* Bilateral or previous proximal humerus fractures on either side
* Splitting fracture of the humeral head or humeral head impression fracture
* Cuff-arthropathy of the contra- or ipsilateral proximal humerus
* Associated nerve or vessel injury
* Any known clotting disorders, severe cardiac and/or pulmonary insufficiency
* Known hypersensitivity or allergy to any of the components of Traumacem V+ Cement Kit
* Any severe systemic disease: class 4 - 6 of the American Society of Anesthesiologists (ASA) physical status classification
* Any not medically managed severe systemic disease: class 3 of the ASA physical status classification
* Recent history of substance abuse (i.e. recreational drugs, alcohol) that would preclude reliable assessment
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Intraoperative Exclusion Criteria:

* Intraoperative decision to use implants other than PHILOS/PHILOS Screw Augmentation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Any occurrence of radiographically confirmed mechanical failure during the first year after treatment. | one year
  Mechanical failures are defined as loss of reduction (≥ 15° increase of varus malposition between the immediate postoperative position and follow-up radiograph, relative change [5 mm] of greater or lesser tuberosity compared to the immediate postoperative position), head impaction (≥ 5 mm difference in outer plate edge and tangent of humeral head between immediate post-op and follow-up. The tangent is determined perpendicular to the humeral neck), screw/plate loosening (any change outwards of screw position in relation to immediate postoperative position) and secondary screw perforation (perforation of one or more screws through the humeral head into the joint space on the follow-up radiograph(and lack of screw perforation on the intra- or postoperative Rx based on a baseline anteroposterior and axial Rx.

SECONDARY OUTCOMES:
Patient reported outcome (Quality of life) | Preoperative, 6 weeks ±7 days, 12 weeks ± 14 days, 6 months ± 30 days, 12 months up to 425 days after surgery
  EuroQol-5D (EQ-5D).
Intra- and postoperative adverse events related to the procedure and/or device | Up to one year
  Implant/surgery , Bone/fracture, Soft tissue of the musculoskeletal system, Wound/other local tissue, Systemic/rest of the body.
Reoperation rate | Up to one year
Surgical details | Intraoperative
  Surgery duration (skin to skin in min).
Description of augmentation details | Intraoperative
  Number of screws augmented.
Surgical details | Intraoperative
  Time of day of surgery.
Surgical details | Intraoperative
  Number and position of screws used.
Surgical details | Intra- /postoperative
  Anatomic/non-anatomic reduction.
Surgical details | Intra- /postoperative
  Restoration of medial support.
Description of augmentation details | Intraoperative
  Number of incidences of direct contrast fluid leakage.
Description of augmentation details | Intraoperative
  Augmentation-related adverse events and their association with fracture characteristics.
Description of augmentation details | Intraoperative
  Volume of injected cement (in ml).
Shoulder function | Preoperative, 6 weeks ±7 days, 12 weeks ± 14 days, 6 months ± 30 days, 12 months up to 425 days after surgery
  Shoulder Pain and Disability Index (SPADI).
Shoulder function | Preoperative, 6 weeks ±7 days, 12 weeks ± 14 days, 6 months ± 30 days, 12 months up to 425 days after surgery
  Constant score.
Shoulder function | Preoperative, 6 weeks ±7 days, 12 weeks ± 14 days, 6 months ± 30 days, 12 months up to 425 days after surgery
  Disabilities of the Arm, Shoulder and Hand Score (QuickDASH).
Relation of patient factors on mechanical failures | Up to one year
  Comorbidity.
Relation of patient factors on mechanical failures | Up to one year
  Mental health with Mini Mental State Examination (MMSE).
Relation of patient factors on mechanical failures | Up to one year
  Bone mineral density (BMD) measured with CT.
Relation of fracture characteristics on mechanical failures | Up to one year
  Number of fracture parts.
Relation of fracture characteristics on mechanical failures | Up to one year
  Severity of displacement.
Relation of fracture characteristics on mechanical failures | Up to one year
  Varus/valgus.
Relation of surgical factors on mechanical failures | Up to one year
  Anatomic/non-anatomic reduction (varus, anteversion etc.).
Relation of surgical factors on mechanical failures | Up to one year
  Restoration of medial support.
Relation of surgical factors on mechanical failures | Up to one year
  Time of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Faeh, Study Director — AO Clinical Investigation and Documentation, Davos, Switzerland; Franz Kralinger, PD, MD, Principal Investigator — Medical University of Innsbruck, Austria
Locations (9):
- Medical University of Innsbruck, Innsbruck, Austria
- UZ Leuven, Leuven, Belgium
- Germany (5):
  - University Hospital RWTH Aachen, Aachen
  - University Medical Center Freiburg, Freiburg im Breisgau
  - Saarland University Medical Center, Homburg
  - BG Clinic Ludwigshafen, Ludwigshafen
  - BG Clinic Tübingen, Tübingen
- Switzerland (2):
  - Cantonal Hospital Lucerne, Lucerne
  - Triemli hospital, Zurich

REFERENCES:
- [Result] Hengg C, Nijs S, Klopfer T, Jaeger M, Platz A, Pohlemann T, Babst R, Franke J, Kralinger F. Cement augmentation of the proximal humerus internal locking system in elderly patients: a multicenter randomized controlled trial. Arch Orthop Trauma Surg. 2019 Jul;139(7):927-942. doi: 10.1007/s00402-019-03142-6. Epub 2019 Feb 25. PMID 30805708
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196
- See also: Link to publication — https://link.springer.com/article/10.1007%2Fs00402-019-03142-6